CLINICAL TRIAL: NCT01003496
Title: Comparing Acute and Continuous Drug Abuse Treatment: A Randomized Clinical Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wright State University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Maryhaven (Unknown); University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIDA/NIH 1RC1DA028467-01; 1RC1DA028467-01 (NIH)
Record Dates: First submitted 2009-10-27; First posted 2009-10-28 (Estimated); Last update posted 2022-03-09 (Actual); Status verified 2022-02

CONDITIONS: Drug Addiction
Keywords: Cocaine; crack; heroin; non-prescribed opioids; contingency management; community reinforcement approach; facilitated therapeutic alliance; chronic disease treatment models
MeSH Terms: conditions — Substance-Related Disorders | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment as Usual (TAU) (Active Comparator)
  Interventions: Behavioral: Treatment as Usual (TAU)
- TAU + Long-Term Recovery Management (LTRM) (Experimental)
  Interventions: Behavioral: TAU + Long-Term Recovery Management

INTERVENTIONS:
Behavioral: Treatment as Usual (TAU) — Outpatient substance abuse treatment
  Arms: Treatment as Usual (TAU)
Behavioral: TAU + Long-Term Recovery Management — Long-Term Recovery Management (LTRM) combines 3 established treatment techniques (Community Reinforcement Approach, Contingency Management, and Facilitated Therapeutic Alliance), each with demonstrated efficacy, into a chronic disease model. In addition, patient cases are kept open, thereby removing potential obstacles to re-engagement with stepped-up care, when indicated. Patients randomly assigned to LTRM will be asked to participate in group sessions each month for 12 months.
  Arms: TAU + Long-Term Recovery Management (LTRM)

SUMMARY:
The purpose of this 2 year study is to conduct a fully powered effectiveness trial comparing recovery trajectories of 200 drug dependent adults (the subjects) who will be randomly assigned to Treatment as Usual (TAU) or TAU + Long-Term Recovery Management (LTRM).

DETAILED DESCRIPTION:
Drug addiction is a chronic illness characterized by problematic drug use, followed by periods of abstinence, reductions in use, or return to problematic drug use. Despite this, substance abuse treatment has traditionally been based on an acute care model. The field needs an addiction management model for drug-dependent patients, which, like disease management for other chronic conditions, provides: 1) initial stabilization; 2) ongoing treatment to maintain clinical gains; 3) monitoring of patient symptoms; and 4) adjustments to the treatment based on the patient's response.

In response to these needs we have developed the Long Term Recovery Management (LTRM) model. LTRM is predicated on initiating long-term addiction management at the onset of substance abuse treatment, extending the length of treatment, expediting the transitions between intensive treatment and maintenance of behavioral change, adapting treatment intensity to patient's response to treatment, and actively facilitating the therapeutic alliance. LTRM combines 3 established treatment techniques (Community Reinforcement Approach, Contingency Management, and Facilitated Therapeutic Alliance), each with demonstrated efficacy, into a chronic disease model. In addition, patient cases are kept open, thereby removing potential obstacles to re-engagement with stepped-up care, when indicated. The LTRM model emphasizes: engagement in continuous long-term treatment and recovery support, therapeutic alliance, and early re-intervention as the main mechanisms for maintenance of behavioral change.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for the study, a subject must:

* At least 18 years of age
* Meet current dependence criteria for stimulants (cocaine/other), opioids (heroin/other), and/or alcohol (if also dependent on cocaine or opioids). Persons who are opioid dependent are eligible if they are not in methadone maintenance therapy; they will be eligible if they are in short-term buprenorphine detoxification
* Self-report use of a primary drug of dependence in the past 60 days; 4) be admitted to outpatient care at Maryhaven
* Willing to participate in the protocol (i.e., to be randomized to treatment condition and agree to attend regular treatment sessions).

Exclusion Criteria:

* Potential subjects will be excluded if they: 1) present with current suicide risk
* Have a current, untreated psychotic disorder
* Plan to relocate outside of the area within 12 months
* Have been sentenced to incarceration of more than 30 days over the next 6 months
* Are alcohol dependent without current dependence on cocaine or opioids.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2009-11-05 (Actual); Primary Completion 2011-07-27 (Actual); Study Completion 2011-07-27 (Actual)

PRIMARY OUTCOMES:
The main outcome is weeks of abstinence from the primary drug of dependence. | 12 months

SECONDARY OUTCOMES:
Secondary outcomes include drug-free days and reduction in HIV risk behaviors. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Robert G Carlson, Ph.D., Principal Investigator — Wright State University Boonshoft School of Medicine; Russel Falck, MA, Study Director — Wright State University Boonshoft School of Medicine; Gregory Brigham, Ph.D., Study Director — Maryhaven; Brenda M Booth, Ph.D., Study Director — University of Arkansas
Locations (1):
- Maryhaven, Columbus, Ohio, United States